CLINICAL TRIAL: NCT06733415
Title: Changes in Energy Expenditure (EE) in Transsexuals Undergoing Hormonal Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0697-22; 0697-22 (Registry Identifier: Changes in Energy Expenditure (EE) in Transsexuals undergoing Hormonal Therapy)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Transgender; Transgender Persons, M01.777.500
Keywords: trangender, metabolic rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CBC, cortisol, glucose, HBA1C , FULL CHEMISTRY, LIPID PANEL, LH FSH ESTRADIOL TESTOSTERONE, PROLACTIN, PROGESTERONE
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Examining Metabolic Rate in Transgender individuals before starting hormonal treatment and 6-12 months after initiation

DETAILED DESCRIPTION:
Study Objective

1. To assess energy expenditure including: resting energy expenditure (RER), - in transgender subjects undergoing hormonal gender affirming treatment.
2. To assess change in Physical Activity (PA) before and after treatment. Methods Study design: A pilot observational prospective study, recruiting 20 transsexuals: 10 transwomen (TW) and 10 transmen (TM).

Criteria for inclusion

1. TW and TM with no prior hormonal therapy in the last one year.
2. Stable weight in last six months (<±5% weight change),

Criteria for exclusion

1. Postmenopausal TM.
2. Oral contraceptive use.
3. Pregnancy or breastfeeding.
4. Glucocorticosteroid treatment
5. Uncontrolled thyroid disorders
6. Use of drugs that potentially impact body metabolism Follow up will be for 6 months.

Baseline tests and after 3 and 6 months of treatment:

1. Anthropometrics:

   1. Body weight will be measured to the nearest 10 g on a digital scale (Seca, 'mBCA') after 12 hours of overnight fast.
   2. Height will be measured with a wireless digital stadiometer (Seca 274) to the nearest 0.1 cm at baseline.
   3. Changes in body composition, including Fat and Fat Free Mass, will be evaluated by multi-frequency bioelectrical impedance analysis (BIA) after 12 hours fasting, using the 'mBCA' body composition analyzer.
   4. Waist and hip circumference will be measured with a tape measure
   5. Resting blood pressure - diastolic and systolic, and heart rate will be measured by a completely automated device (Omron, M7) after sitting at least 10 min without distractions (e.g. cell phones).

   Body weight, waist and hip circumference, body composition, blood pressure and resting heart rate measurements will be made pre and 3, 6 months post therapy.
2. Fasting (12 hours) blood tests pre and post therapy: (Blood tests will take place in the endocrinology institute in Ichilov hospital.)

   1. Hormone analysis: TSH T4FREE T3, CORTISOL LH FSH ESTRADIOL PROGESTERONE, testosterone, bioavailable testosterone, DHEAS
   2. Clinical chemistry: electrolytes, kidney function tests, liver function tests
   3. Complete blood count
   4. Lipid profile
   5. Glucose and HbA1c-levels, INSULIN
3. Fecal microbiota pre and post therapy
4. Measurement of REE will be measured over a 60-minute period using whole-room indirect calorimeter (WRIC) Participants will enter the WRIC at 7am after overnight 12 hours of fasting and at least 24 hours after the last bout of any structured exercise, with instructions to avoid unnecessary activity on the morning of testing, . They will then be instructed to maintain a supine position until 8pm for measuring REE.
5. Changes in daily physical activity and sedentary behavior will be assessed for 7 days pre- and post- hormonal therapy by a tri-axial accelerometer (ActiGraph GT9X Link, Pensacola, Florida).

Whole human room calorimetry The REE will be measured by indirect calorimetry in a small WRIC (~11,500 liters) pre and post hormonal therapy. Air in the calorimeter will be removed at 240 L/min. Oxygen uptake and carbon dioxide production will be measured using gas analyzers (Promethion room calorimeter systems) and calculated by ExpeData software (Sable Systems, USA). The O2 and CO2 gas analyzers will be calibrated using dry chemicals before each experiment, and once a week by using standardized gas mixtures. To calculate EE we will use the Weir's equation (EE = 3.9 × VO2 (L) + 1.1 × VCO2 (L)) and the respiratory quotient (RQ) will be calculated as VCO2/VO2. The accuracy of the WRIC for the measurement of EE, determined repeatedly using a 3 hours N2 injection test, was 99.4% ± 2.6% for O2 consumption. For the duration of the test, the participant will be asked to remain motionless and awake in a supine position, lightly clothed in a thermoneutral (22°C-23°C), dimly lit and quiet room.

Statistical Analysis We plan on using two-tailed tests in SAS with α=0.05. Power analysis indicates that 10 individuals will be needed to have 80% power to detect an 80 kcal/day difference in 24-hr energy expenditure (the primary endpoint), based on unpublished data indicating a within-subjects standard deviation of σ=79 kcal/day (Ravussin et al. 2019). Baseline data and the data for each arm will be reported in the text as raw mean ± SD, while the treatment effects or differences between arms (denoted Δ) are reported as least squares mean ± SEM. The treatment effects and associated p-values were computed using linear mixed models with heterogeneous compound symmetry, with participants as the random effect and the treatment, period, sequence, and BMI as fixed effects, using the Satterthwaite method for calculating degrees of freedom.

ELIGIBILITY:
Inclusion Criteria:

1. TW and TM with no prior hormonal therapy in the last one year. 2. Stable weight in last six months (<±5% weight change),

-

Exclusion Criteria:

1. Postmenopausal TM.
2. Oral contraceptive use.
3. Pregnancy or breastfeeding.
4. Glucocorticosteroid treatment
5. Uncontrolled thyroid disorders
6. Use of drugs that potentially impact body metabolism

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Transgender individuals prior to gender affirming hormonal therapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
RESTING METABOLIC RATE | 6-12 months
  Methods Study design: A pilot observational prospective study, recruiting 34 transsexuals: 17 transwomen (TW) and 17 transmen (TM).
  Criteria for inclusion
  1. TW and TM with no prior hormonal therapy in the last one year.
  2. Stable weight in last six months (<±5% weight change),
  Criteria for exclusion
  1. Postmenopausal TM.
  2. Oral contraceptive use.
  3. Pregnancy or breastfeeding.
  4. Glucocorticosteroid treatment
  5. Uncontrolled thyroid disorders
  6. Use of drugs that potentially impact body metabolism Follow up will be for 6 months.
  Baseline tests and after 3 and 6 months of treatment:
  1. Anthropometrics:
  1. Body weight will be measured to the nearest 10 g on a digital scale (Seca, 'mBCA') after 12 hours of overnight fast.
  2. Height will be measured with a wireless digital stadiometer (Seca 274) to the nearest 0.1 cm at baseline.
  3. Changes in body composition, including Fat and Fat Free Mass, will be evaluated by multi-frequency bioelectrical impedance analysis (BIA) after 12 hour

CONTACTS AND LOCATIONS:
Overall Officials: Yael Sofer, MD, Principal Investigator — Department of Endocrinology, Metabolism and Hypertension, Tel Aviv Sourasky Medical Center and Tel Aviv University
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided
As I have not requested a permission for this from the local ethics committee I cannot promise to share.